CLINICAL TRIAL: NCT05979922
Title: Mindfulness-based Cognitive Coping Mobile App Intervention for Caregivers of Individuals With Alzheimer's Disease
Brief Title: Mindfulness-based Cognitive Coping for ADRD Caregivers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Photozig, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pz-A108a; R44AG058277 (NIH)
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Caregiver Stress
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caring Mind mobile app (Experimental): Participants will receive the Caring Mind mobile app containing the Mindfulness-based Cognitive Coping program.
  Interventions: Behavioral: Mindfulness-based Cognitive Coping
- Traditional educational program (Active Comparator): Participants will receive a traditional educational/resources program, containing a downloadable workbook and online resources.
  Interventions: Behavioral: Traditional Educational/Resources Program

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Coping — Participants will receive the Caring Mind mobile app containing the Mindfulness-based Cognitive Coping program.
  Arms: Caring Mind mobile app
Behavioral: Traditional Educational/Resources Program — Participants will receive a traditional educational/resources program, containing a downloadable workbook and online resources.
  Arms: Traditional educational program

SUMMARY:
This project will evaluate the effectiveness of the Mindfulness-based Cognitive Coping (MCC) intervention to alleviate stress and depressive symptoms of caregivers of Individuals with Alzheimer's Disease and Related Dementia.

ELIGIBILITY:
Inclusion Criteria:

* Care for an individual with Alzheimer's Disease or Related Dementia (ADRD).
* Own a smartphone or tablet and have Internet access.
* Minimum age of 18 years old.
* Able to read and speak English.
* Spend at least 8 hours/week caring for a person with dementia.
* Plan to stay in the area for six months.

Exclusion Criteria:

* Severe psychological or physical illness.
* Cognitive impairment or any serious medical problem that interferes with caregiving role.
* Caring for ADRD patient with a life expectancy less than six months.
* Unwillingness to participate in all aspects of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Photozig, Inc., Campbell, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Caring Mind Mobile App | Traditional Educational Program
Started | 88 | 86
Completed | 59 | 58
Not Completed | 29 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caring Mind Mobile App | Traditional Educational Program | Total
Number analyzed (Participants) | 88 | 86 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (11.8) | 58.1 (9.4) | 57.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 79 | 158
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 83 | 81 | 164
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Center for Epidemiological Studies Depression Scale
Description: The Center for Epidemiological Studies Depression scale (CES-D) is a 20-item measure that asks about the frequency of depressive symptoms (affective, psychological, and somatic) within the past week.The scale refers to the caregiver. Minimum score (best value)=0. Maximum score (worst value)=60. Higher values represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caring Mind Mobile App | Traditional Educational Program
Number analyzed (Participants) | 59 | 58
score on a scale | 17.1 (9.66) | 21.98 (12.48)

2. Primary Outcome: Perceived Stress Scale
Description: The "Perceived Stress Scale" measures the overall level of stress. This instrument contains 10 items accessing overall appraisals of stress in the past month. The scale refers to the caregiver. Minimum score (best value)=0. Maximum score (worst value)=40. Higher values represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caring Mind Mobile App | Traditional Educational Program
Number analyzed (Participants) | 59 | 58
score on a scale | 17.12 (7.58) | 19.38 (6.97)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Definitions are the same as the ones from clinicaltrials.gov.
Arm/Group | Caring Mind Mobile App | Traditional Educational Program
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/86
Other Adverse Events (participants affected / at risk) | 0/88 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT05979922/Prot_SAP_000.pdf